CLINICAL TRIAL: NCT06746181
Title: Effect of Different Inspired Oxygen Concentrations on Intraoperative Recruitment Outcomes in Patients Undergoing Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Ju Gao, Study Director, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024ky310
Record Dates: First submitted 2024-12-17; First posted 2024-12-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Atelectasis, Postoperative
Keywords: Inhaled oxygen concentration; lung recruitment
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A: FiO2 = 30% (Experimental): FiO2 of group A = 30%. If SPO2 < 94%, improve FiO2; if FiO2≥40%, eliminate the patient.
  Interventions: Behavioral: Fraction of inspiration O2(FiO2)
- B: FiO2＝40% (Experimental): FiO2＝40%
  Interventions: Behavioral: Fraction of inspiration O2(FiO2)
- C: FiO2＝60% (Experimental): FiO2＝60%
  Interventions: Behavioral: Fraction of inspiration O2(FiO2)
- D: FiO2＝80% (Experimental): FiO2＝80%
  Interventions: Behavioral: Fraction of inspiration O2(FiO2)

INTERVENTIONS:
Behavioral: Fraction of inspiration O2(FiO2) — After the patient was admitted to the room, anesthesia induction was performed after pre-oxygenation for 3 minutes. Tracheal intubation was carried out once the medication had fully taken effect. After the surgery began, the inspired oxygen concentration was adjusted for each group. The first lung recruitment maneuver was performed 10 minutes later, and subsequent lung recruitment maneuvers were conducted when pulmonary compliance returned to baseline levels. This process was repeated, with all patients undergoing one final lung recruitment maneuver immediately at the end of the surgery.

SUMMARY:
This study intends to evaluate the effect of different inhaled oxygen concentrations on the effect of lung recruitment in patients undergoing abdominal surgery. During perioperative mechanical ventilation, higher FiO2 is usually given to prevent the occurrence of hypoxemia, but there are no conclusions about the setting of optimal FiO2 during surgery.

Dynamic pulmonary compliance enables real-time monitoring of alveolar changes and is used to assess pulmonary function in intraoperative patients. The value of compliance represents the number of air-containing alveoli; the more alveoli are trapped, the less air-containing tissue there is and the lower the compliance. Lung recruitment, as part of a lung-protective ventilation strategy, is effective in opening alveoli and improving oxygenation. This single-center, randomized controlled trial will explore the optimal inspired oxygen concentration that allows patients to benefit from lung recruitment and the duration of improvement in lung compliance after lung recruitment.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status classification: I or II.
* Adults aged 18 to 64 years, regardless of gender.
* BMI between 18 kg/m² and 25 kg/m².
* Patients undergoing elective abdominal surgery under general anesthesia.
* Patients with estimated operating time ≥1.5h and intraoperative bleeding ≤500ml.
* Patients who have provided written informed consent after understanding the study purpose, procedures, and potential risks.

Exclusion Criteria:

* Previous thoracic surgery.
* Chest X-ray or CT suggestive of pneumothorax or alveoli.
* Lung disease: chronic bronchitis, asthma, moderate to severe obstructive ventilatory dysfunction.
* Preoperative pulse oxygen saturation (SpO2) <90% on breathing air or SpO2 <95% on oxygen.
* Contraindications to lung reanimation: high intracranial pressure, hypovolemic shock, right heart failure.
* Severe heart disease (New York Heart Association, NYHA class III or IV.
* Acute coronary syndrome or sustained ventricular tachyarrhythmia).
* Participation in other interventional studies or refusal of enrollment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Duration of improvement in lung compliance | during the surgery
  Time to return to baseline levels of lung compliance after lung recruitment

SECONDARY OUTCOMES:
Incidence of hypoxemia during PACU | From the time of entry to the PACU to the time of exit from the PACU
Incidence of pulmonary atelectasis at the end of surgery | Surgery complete, extubation immediate
Incidence of pulmonary complications within 3 days after surgery | From the end of surgery to 3 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared. Data will include demographic characteristics, procedural details, and outcome measures. Access will be granted to qualified researchers upon request via a secure data repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified individual participant data (IPD) will be available starting 6 months after the publication of the primary study results. Data will remain available for 3 years.
Access Criteria: Qualified researchers affiliated with academic, governmental, or non-profit institutions may request access to the IPD. Requests must include a detailed research proposal, institutional review board (IRB) approval (if applicable), and a signed data-sharing agreement. Access will be provided to de-identified data relevant to the study objectives, including demographic information, procedural details, and primary/secondary outcome measures. Data will be shared via a secure repository upon approval of the request.

REFERENCES:
- [Result] Edmark L, Ostberg E, Scheer H, Wallquist W, Hedenstierna G, Zetterstrom H. Preserved oxygenation in obese patients receiving protective ventilation during laparoscopic surgery: a randomized controlled study. Acta Anaesthesiol Scand. 2016 Jan;60(1):26-35. doi: 10.1111/aas.12588. Epub 2015 Aug 3. PMID 26235391
- [Result] Andrade FSRM, Ambrosio AM, Rodrigues RR, Facco LL, Goncalves LA, Garcia Filho SG, Dos Santos RT, Rossetto TC, Pereira MAA, Fantoni DT. The optimal PEEP after alveolar recruitment maneuver assessed by electrical impedance tomography in healthy horses. Front Vet Sci. 2022 Dec 9;9:1024088. doi: 10.3389/fvets.2022.1024088. eCollection 2022. PMID 36570501
- [Result] Lee JH, Choi S, Ji SH, Jang YE, Kim EH, Kim HS, Kim JT. Effect of an ultrasound-guided lung recruitment manoeuvre on postoperative atelectasis in children: A randomised controlled trial. Eur J Anaesthesiol. 2020 Aug;37(8):719-727. doi: 10.1097/EJA.0000000000001175. PMID 32068572
- [Result] Wu XZ, Xia HM, Zhang P, Li L, Hu QH, Guo SP, Li TY. Effects of ultrasound-guided alveolar recruitment manoeuvres compared with sustained inflation or no recruitment manoeuvres on atelectasis in laparoscopic gynaecological surgery as assessed by ultrasonography: a randomized clinical trial. BMC Anesthesiol. 2022 Aug 16;22(1):261. doi: 10.1186/s12871-022-01798-z. PMID 35974310
- [Result] Neira VM, Kovesi T, Guerra L, Campos M, Barrowman N, Splinter WM. The impact of pneumoperitoneum and Trendelenburg positioning on respiratory system mechanics during laparoscopic pelvic surgery in children: a prospective observational study. Can J Anaesth. 2015 Jul;62(7):798-806. doi: 10.1007/s12630-015-0369-0. Epub 2015 Apr 23. PMID 25902890
- [Result] Young CC, Harris EM, Vacchiano C, Bodnar S, Bukowy B, Elliott RRD, Migliarese J, Ragains C, Trethewey B, Woodward A, Gama de Abreu M, Girard M, Futier E, Mulier JP, Pelosi P, Sprung J. Lung-protective ventilation for the surgical patient: international expert panel-based consensus recommendations. Br J Anaesth. 2019 Dec;123(6):898-913. doi: 10.1016/j.bja.2019.08.017. Epub 2019 Oct 3. PMID 31587835

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT06746181/Prot_ICF_000.pdf